CLINICAL TRIAL: NCT05731947
Title: A Phase 1/2 Study to Investigate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Efficacy of SNDX-5613 in Patients With Colorectal Cancer and Other Solid Tumors
Brief Title: Evaluation of Revumenib in Participants With Colorectal Cancer and Other Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Syndax Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SNDX-5613-0706
Expanded Access: NCT05918913 (No longer available)
Record Dates: First submitted 2023-02-07; First posted 2023-02-16 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Colorectal Cancer; Solid Tumors
Keywords: SNDX-5613; Revumenib; Menin
MeSH Terms: conditions — Colorectal Neoplasms | interventions — revumenib; Drug Therapy

STUDY DESIGN:
Intervention Model Description: Phase 1a dose escalation portion of the study will employ a Rolling 6 trial design, followed by a Phase 1b signal-seeking portion, and a Phase 2 randomized (2:1) signal confirmation portion.
  Phase 1: Non-randomized; Phase 2: Randomized
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase 1a: Dose Escalation (Experimental): Participants will receive revumenib tablets or capsules three times a day (TID) or two times a day (BID) from Day 1 of each 28-day cycle.
  Interventions: Drug: Revumenib
- Phase 1b: Signal-Seeking (Experimental): Participants will receive revumenib tablets TID or BID from Day 1 of each 28-day cycle.
  Interventions: Drug: Revumenib
- Phase 2: Revumenib (Experimental): Participants will receive revumenib tablets TID or BID from Day 1 of each 28-day cycle.
  Interventions: Drug: Revumenib
- Phase 2: Chemotherapy (Active Comparator): Participants will receive chemotherapy from Day 1 of each 28-day cycle.
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: Revumenib — Revumenib administered orally with or without food. Participants may continue to receive treatment until disease progression or until they experience unacceptable toxicity.
  Other Names: SNDX-5613
  Arms: Phase 1a: Dose Escalation; Phase 1b: Signal-Seeking; Phase 2: Revumenib
Drug: Chemotherapy — Either Lonsurf® or Stivarga® administered per the investigator's choice at the respective drug label's dose and schedule. Participants may continue to receive treatment until disease progression or until they experience unacceptable toxicity.
  Arms: Phase 2: Chemotherapy

SUMMARY:
This study will evaluate the safety, tolerability, pharmacokinetics (PK), and anti-tumor activity of revumenib in participants with colorectal cancer (CRC) or other solid tumors who have failed at least 1 prior line of therapy.

DETAILED DESCRIPTION:
The study will be conducted in two parts. The Phase 1 portion of the study consists of a dose escalation cohort, and a signal-seeking expansion where anti-tumor activity signals will be evaluated. The Phase 2 portion of the study will further confirm the anti-tumor activity signals of revumenib.

ELIGIBILITY:
Key Inclusion Criteria:

* Male and female participants aged ≥18 years
* Participants with metastatic CRC or other solid tumors
* Evidence of locally recurrent or metastatic disease based on imaging studies within 28 days of cycle 1/day 1 (C1D1)
* CRC participants must have had at least one line of standard-of-care therapy and must have progressed on or been intolerant to, or unable to receive oxaliplatin, irinotecan, and bevacizumab in the advanced/metastatic setting.
* Other solid tumor participants must have had all approved standard therapies that are available to the participant, unless contraindicated or intolerable.
* Participants must have experienced documented unequivocal progressive disease by either RECIST v1.1 or clinical assessment, or experienced unacceptable toxicity with their prior therapy.
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 to 1
* If receiving radiation therapy, has had a 2-week washout period following completion of the treatment prior to receiving the C1D1 dose and continues to have at least 1 measurable lesion
* At least 42 days since prior immunotherapy, including tumor vaccines and checkpoint inhibitors, and at least 21 days since receipt of chimeric antigen receptor therapy or other modified T-cell therapy
* Adequate bone marrow, renal, cardiac, and liver function

Key Exclusion Criteria:

* Participant has a prior history of malignant bowel obstruction requiring hospitalization in the 6 months prior to enrollment
* Participant has a history of uncontrolled ascites, defined as symptomatic ascites and/or repeated paracenteses for symptom control in the past 3 months
* Detectable human immunodeficiency virus (HIV) viral load within the previous 6 months. Participants with a known history of HIV 1/2 antibodies must have viral load testing prior to study enrollment
* Hepatitis B and/or C
* Any of the following within the 6 months prior to study entry: myocardial infarction, uncontrolled/unstable angina, congestive heart failure (New York Heart Association Classification Class ≥II), life-threatening, uncontrolled arrhythmia, cerebrovascular accident, or transient ischemic attack
* Corrected QT interval (QTc) >450 milliseconds
* Any gastrointestinal (GI) issue of the upper GI tract likely to affect oral drug absorption or ingestion (for example, gastric bypass, gastroparesis)
* Cirrhosis with a Child-Pugh score of B or C
* Brain metastasis except for those participants who have completed definitive therapy, are not on steroids, have a stable neurologic status for at least 4 weeks after completion of the definitive therapy and steroids, and do not have neurologic dysfunction that would confound the evaluation of neurologic and other adverse events (AEs)
* History of or any concurrent condition, therapy, laboratory abnormality, or allergy to excipients that in the Investigator's opinion might confound the results of the study, interfere with the participant's ability to participate for the full duration of the study, or not be in the best interest of the participant to participate
* Participant has received prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study baseline or who has not recovered (that is, ≤Grade 1 or at baseline) from AEs related to a previously administered agent.
* Participation in another therapeutic interventional clinical study in which an investigational agent was administered within 30 days before starting revumenib
* Participant has received a transfusion of blood products or administration of colony stimulating factors within 4 weeks of the first dose of the study drug
* History of additional malignancy within the prior 5 years, excluding adequately treated basal cell carcinoma, squamous cell of the skin, cervical intraepithelial neoplasia/cervical carcinoma in situ, or melanoma in situ or ductal carcinoma in situ of the breast

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2023-04-04 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Phase 1a: Number of Participants Experiencing Dose Limiting Toxicities | Up to Day 29
Phase 1: Number of Participants Experiencing Treatment-emergent Adverse Events (TEAEs) | Approximately 12 months
Phase 1b: Disease Control Rate (DCR) | Approximately 6 months
Phase 1b: Overall Response Rate (ORR) | Approximately 6 months
Phase 2: Progression Free Survival (PFS) | Approximately 4 months

SECONDARY OUTCOMES:
Phase 1: Maximum Plasma Concentration (Cmax) of Revumenib | Predose up to approximately 12 months
Phase 1: Time to Maximum Plasma Concentration (Tmax) of Revumenib | Predose up to approximately 12 months
Phase 1: Area Under the Plasma Concentration Versus Time Curve (AUC) of Revumenib | Predose up to approximately 12 months
Phase 2: AUC of Revumenib | Predose up to approximately 6 months
Phase 2: Cmax of Revumenib | Predose up to approximately 6 months
Phase 2: Tmax of Revumenib | Predose up to approximately 6 months
Phase 2: Number of Participants Experiencing TEAEs | Approximately 3 years
Phase 2: Overall Survival (OS) | Approximately 5 years
Phase 2: DCR at 6 Cycles (28-Day Cycles) as Assessed by Blinded Radiographic Review | Approximately 6 months
Phase 2: ORR as Assessed by Blinded Radiographic Review Using Response Evaluation Criteria in Solid Tumors (RECIST), version (v)1.1 | Approximately 6 months
Phase 2: Duration of Response (DOR) as Assessed by Blinded Radiographic Review | Approximately 3 years
Phase 2: DCR at 6 Cycles (28-Day Cycles) as Assessed by the Investigator | Approximately 6 months
Phase 2: ORR as Assessed by the Investigator per RECIST v1.1 | Approximately 6 months
Phase 2: DOR as Assessed by the Investigator | Approximately 3 years

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Honor Health Research Institute, Scottsdale, Arizona
  - Massachusetts General Hospital, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, Manhattan, New York
  - Gabrail Cancer Center, Canton, Ohio
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Inova Schar Cancer Institute, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No